CLINICAL TRIAL: NCT05256290
Title: A Phase 1/2 Study to Assess BDTX-1535, an Oral EGFR Inhibitor, in Patients With Glioblastoma or Non-Small Cell Lung Cancer
Brief Title: Phase 1/2 Study of Silevertinib (BDTX-1535) in Patients With Glioblastoma or Non-Small Cell Lung Cancer With EGFR Mutations
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Black Diamond Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BDTX-1535-101
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer; Advanced Non-Small Cell Squamous Lung Cancer; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Lung Cancer; NSCLC; Advanced Lung Carcinoma; Epidermal Growth Factor Receptor C797S; Epidermal Growth Factor Receptor G719X; EGF-R Positive Non-Small Cell Lung Cancer; EGFR-TKI Resistant Mutation
Keywords: EGFR alterations; EGFR L858R; EGFR Exon 19 del; EGFR inhibitor; intrinsic resistance NSCLC EGFR; acquired resistance NSCLC EGFR; intracranial disease; brain metastases; central nervous system metastases; CNS metastases; uncommon NSCLC EGFR mutations; C797S acquired resistance EGFR mutation; non-classical NSCLC EGFR mutations; classical NSCLC EGFR mutations; EGFR PACC NSCLC mutations; EGFR E709A/G/K/Q/V; EGFR E709_T710delinsD/T; EGFR G719A/C/D/R/S; EGFR G724S; EGFR L718Q/V; EGFR L747S/P, L747_A750delinsP, L747_P753delinsS; Second-site EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Dose Escalation - Monotherapy (Recruitment Closed) (Experimental): * Advanced/metastatic NSCLC with acquired resistance EGFR mutation (eg, C797S), following a 3rd generation EGFR inhibitor in the 1st line setting (in the absence of concurrent T790M).
  * Advanced/metastatic NSCLC with non-classical EGFR mutation (eg, G719X) following standard-of-care therapy with an EGFR inhibitor
  * Recurrent GBM with confirmed EGFR alterations (including amplification, mutation, and/or variant)
  Interventions: Drug: silevertinib (BDTX-1535) monotherapy
- Phase 2 Cohort 1: NSCLC EGFR Non-Classical Driver Mutations (Experimental): Advanced/metastatic NSCLC with a non-classical driver EGFR mutation following up to 2 lines of therapy with only 1 prior EGFR targeted regimen (third-generation preferred; other approved EGFR inhibitors acceptable)
  Interventions: Drug: silevertinib (BDTX-1535) monotherapy
- Phase 2 Cohort 2: NSCLC EGFR Acquired Resistance (C797S) Mutation (Experimental): Advanced/metastatic NSCLC with the acquired resistance C797S EGFR mutation following up to 2 lines of therapy, including only 1 EGFR targeted regimen, which must be a third generation EGFR TKI (eg, osimertinib)
  Interventions: Drug: silevertinib (BDTX-1535) monotherapy
- Phase 2 Cohort 3: Treatment Naive NSCLC EGFR Non-Classical Driver Mutations (Experimental): Treatment-naïve (first-line) advanced/metastatic NSCLC with a non-classical driver EGFR mutation (1 cycle of chemotherapy or immune checkpoint inhibitor are permitted). Patients with co-occurring L858R mutations and a non-classical mutation are eligible for inclusion.

INTERVENTIONS:
Drug: silevertinib (BDTX-1535) monotherapy — Silevertinib (BDTX-1535) is a 4th generation irreversible brain penetrant EGFR MasterKey inhibitor, which targets a family of oncogenic EGFR classical and non-classical driver and resistance mutations in NSCLC.
  Arms: Phase 1 Dose Escalation - Monotherapy (Recruitment Closed); Phase 2 Cohort 1: NSCLC EGFR Non-Classical Driver Mutations; Phase 2 Cohort 2: NSCLC EGFR Acquired Resistance (C797S) Mutation

SUMMARY:
BDTX-1535-101 is an open-label, Phase 1 dose escalation and Phase 2 multiple cohort study designed to evaluate the safety, pharmacokinetics (PK), optimal dosage, central nervous system (CNS) activity, and antitumor activity of silevertinib (BDTX-1535). The study population comprises adults with either advanced/metastatic non-small cell lung cancer (NSCLC) with non-classical or acquired epidermal growth factor receptor (EGFR) resistance (EGFR C797S) mutations with or without CNS disease (in Phase 1 and Phase 2), or glioblastoma (GBM) expressing EGFR alterations (Phase 1 only). All patients will self-administer silevertinib (BDTX-1535) monotherapy by mouth in 21-day cycles.

Phase 1 enrollment is now complete. Phase 2 is currently ongoing.

ELIGIBILITY:
Phase 2 Eligibility:

Key Inclusion Criteria Required for locally advanced or metastatic NSCLC:

* Measurable disease by RECIST 1.1 criteria.
* Adequate bone marrow or organ function.
* Life expectancy of ≥ 3 months.
* Sufficient performance status.
* Confirmed NSCLC, without small cell lung cancer transformation with or without brain metastases.
* Disease progression following or intolerance of standard of care (excluding patients in the treatment-naïve non-classical driver cohort):

  * Cohort 1 (Non-Classical driver cohort): Advanced/metastatic NSCLC with a non-classical driver EGFR mutation (eg, G719X) following up to 2 lines of therapy with only 1 prior EGFR TKI regimen (third-generation preferred; other approved EGFR TKI acceptable).
  * Cohort 2 (Acquired resistance C797S cohort): Advanced/metastatic NSCLC with the acquired resistance C797S EGFR mutation following up to 2 lines of therapy, including only one EGFR TKI, which must be a third generation EGFR TKI (eg, osimertinib).
  * Cohort 3 (First-line non-classical driver cohort): Treatment-naïve advanced/metastatic NSCLC with a non-classical driver EGFR mutation (1 cycle of chemotherapy or immune checkpoint inhibitor are permitted). Patients with co-occurring L858R mutations and a non-classical mutation are eligible for inclusion.
* Identification of one (or more) of the following EGFR mutations by Next Generation Sequencing (NGS) as determined by a local assay performed in a validated laboratory in the absence of other known resistance mutations (eg, T790M, MET):

  * Non-classical driver EGFR mutations (eg, L861R, S768I, G719X).
  * EGFR acquired resistance mutation (eg, C797S) to a 3rd generation EGFR TKI.
  * For Phase 2, dose expansion, patients in Cohort 1 who received 3rd generation EGFR TKI (eg, osimertinib), the NGS report within 6 months prior to the start of Screening is acceptable. For patients in Cohort 2, the NGS report must be from the last disease progression on the immediate prior therapy. For patients in Cohort 3, the NGS report must be at the time of diagnosis.

Key Exclusion Criteria:

* Known resistant mutations in tumor tissue or by liquid biopsy (eg, T790M, MET).
* Received more than 1 EGFR TKI therapy (ie, erlotinib or gefitinib) for the treatment of metastatic or recurrent EGFR NSCLC.
* Any history of interstitial lung disease related to EGFR TKI use.
* Symptomatic or radiographic leptomeningeal disease.
* Symptomatic brain metastases or spinal cord compression requiring urgent clinical intervention.
* Unresolved toxicity from prior therapy.
* Significant cardiovascular disease.
* Major surgery within 4 weeks of study entry or planned during study.
* Ongoing or recent anticancer therapy or radiation therapy.
* Evidence of malignancy (other than study-specific malignancies) requiring active therapy within the next 2 years.
* Active hepatitis B or C infection and/or known human immunodeficiency virus (HIV) carrier.
* Poorly controlled gastrointestinal disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Dose Escalation: To determine the maximum tolerated dose (MTD), if one exists, and the preliminary recommended Phase 2 dose(s) (RP2D[s]) of silevertinib (BDTX-1535) | The first treatment 21-day cycle (Cycle 1)
  Dose-limiting toxicities (DLTs) in Cycle 1
Phase 2: To assess antitumor efficacy of silevertinib (BDTX-1535) | Day 1 every 2 cycles starting on Cycle 3 Day 1 to study completion, approximately 1 year (each cycle is 21 days)
  Objective response rate (ORR) as assessed by Investigator using RECIST version 1.1

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Incidence and severity of treatment-emergent adverse events (TEAEs) | Through study completion, approximately 1 year
Phase 1 and Phase 2: To characterize the plasma concentration of silevertinib (BDTX-1535) following single and multiple dosing | Cycle 1 Days 1, 2, 15, and 16, Cycles 2 to 5 Day 1, and Day 1 of every other cycle thereafter to study completion, approximately 1 year (each cycle is 21 days)
Phase 1: To assess the preliminary antitumor activity of silevertinib (BDTX-1535) by objective response as assessed by RECIST version 1.1 (for patients with NSCLC) or Response Assessment in Neuro-oncology (RANO) (for patients with GBM) | Day 1 every 2 cycles starting on Cycle 3 Day 1 to study completion, approximately 1 year (each cycle is 21 days)
Phase 1: To assess the effect of tablet formulation on the plasma concentration of silevertinib (BDTX-1535) | Two timepoints during the first cycle: Cycle 0 (7 days prior to Cycle 1 Day 1) and Cycle 1 Day 1 only (each cycle is 21 days)
Phase 1: To assess the effect of food on the plasma concentration of silevertinib (BDTX-1535) | Two timepoints during the first cycle: Cycle 0 (7 days prior to Cycle 1 Day 1) and Cycle 1 Day 1 only (each cycle is 21 days)
Phase 2: To assess duration of tumor response by RECIST version 1.1 | Day 1 every 2 cycles starting at Cycle 3 Day 1 to study completion, approximately 1 year (each cycle is 21 days)
Phase 2: To assess progression free survival by RECIST version 1.1 | Day 1 every 2 cycles starting at Cycle 3 Day 1 to study completion, approximately 1 year (each cycle is 21 days)
Phase 2: To determine the optimal dosage of silevertinib (BDTX-1535) (100 mg or 200 mg daily dose) | At least the first treatment 21-day cycle (Cycle 1) for select patients enrolled into the Phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Black Diamond Therapeutics, Study Director — Black Diamond Therapeutics
Locations (25):
- United States (25):
  - University of Alabama, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope Huntington Beach, Huntington Beach, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sibley Memorial Hospital Johns Hopkins Medicine, Washington D.C., District of Columbia
  - Mayo Clinic- Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute - Baptist Health South Florida, Miami, Florida
  - UHP- University of Hawaii Cancer Center, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Kansas Cancer Center, Fairway, Kansas
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic- Rochester, Rochester, Minnesota
  - Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Hospitals - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Next Ocology, Fairfax, Virginia
  - Fred Hutchinson Cancer Center/University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No